CLINICAL TRIAL: NCT00955604
Title: Investigation of the Occurrence of Serotonin Toxicity in Parkinson's Disease (PD) Patients Treated Concomitantly With Rasagiline and Antidepressants, Using Retrospective Chart Review
Brief Title: Azilect + Antidepressant Chart Review
Acronym: STACCATO
Status: Completed | Type: Observational
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TVP-1012/PM102 CR
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Serotonin Syndrome
Keywords: Parkinson's Disease; Serotonin Toxicity; Rasagiline; Antidepressants; Chart Review; Retrospective
MeSH Terms: conditions — Serotonin Syndrome; Parkinson Disease | interventions — Antidepressive Agents; rasagiline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group R+AD: Group R+AD Rasagiline and an antidepressant (SRIs, SNRIs, St. John's wort and/or TCAs) for at least 14 days
  Interventions: Drug: Group R+AD Rasagiline + Antidepressant
- Group R: At least 2 months of rasagiline
  Interventions: Drug: Group R Rasagiline
- Group AD: At least 2 months of Anti-PD and Rasagiline
  Interventions: Drug: Group AD Anti-PD + Antidepressant

INTERVENTIONS:
Drug: Group R+AD Rasagiline + Antidepressant — Rasagiline and an antidepressant (SRIs, SNRIs, St. John's wort and/or TCAs) at least 14 days
  Other Names: Azilect
  Groups: Group R+AD
Drug: Group R Rasagiline — At least 2 months of rasagiline
  Other Names: Azilect
  Groups: Group R
Drug: Group AD Anti-PD + Antidepressant — An approved dopaminergic medication for PD. (2 months of treatment with an antidepressant medication.
  Groups: Group AD

SUMMARY:
To identify the occurrence of serotonin toxicity in Parkinson's Disease (PD) patients receiving antidepressant therapy and rasagiline, compared to those receiving rasagiline without antidepressant medications and compared to PD patients receiving antidepressants, but not rasagiline.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with a diagnosis of PD
2. Rasagiline treatment as mono- or adjunct therapy for PD with concomitant antidepressant medication (SSRIs, SNRIs, St. John's wort and/or TCAs) at any time during the specified review period, OR Rasagiline treatment as mono- or adjunct therapy for PD without concomitant antidepressant medication (SSRIs, SNRIs, St. John's wort and/or TCAs) at any time during the specified review period. OR Antidepressant therapy (SSRIs, SNRIs, St. John's wort and/or TCAs) and any other dopaminergic anti-PD treatment besides rasagiline or selegiline at any time during the specified review period
3. Willing to consent to review of office chart and to review of records of ER visits and/or hospitalizations corresponding to the review window, if required
4. Patients previously participating in a rasagiline clinical trial (and their follow-up protocols) are eligible, provided that they did not receive antidepressant therapy during trial participation.
5. In addition to the above criteria, each group has specific inclusion criteria stated below:

   * Group R+AD: Enrollment in this group requires that patients must have taken rasagiline and an antidepressant (SSRIs, SNRIs, St. John's wort and/or TCAs, regardless of indication) within 14 days of each other (or five weeks, if fluoxetine preceded rasagiline).
   * Group R: Enrollment in this group requires patients must have at least 2 months of rasagiline use.
   * Group AD: Patients must be taking an approved dopaminergic medication for PD. Enrollment in this group requires that patients must have at least 2 months of treatment with an antidepressant medication.

Exclusion Criteria:

1. Use of rasagiline for any indication other than PD
2. Patients taking a monoamine oxidase inhibitor (MAOI) antidepressant and/or selegiline
3. Inability or unwillingness to request records of ER visits and/or hospitalizations corresponding to the review period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female patients with a diagnosis of PD:
  * who received rasagiline at any dose, as mono- or adjunct therapy for PD, with concomitant antidepressant medication, OR
  * who received rasagiline at any dose, as mono- or adjunct therapy for PD, without concomitant antidepressant medication, OR
  * who received antidepressant medication and any other dopaminergic anti-PD therapy besides rasagiline or selegiline including dopaminergic agents, anticholinergics, amantadine, deep brain stimulation (DBS), pallidotomy, etc.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The frequency of serotonin toxicity, as determined by the Adjudication Committee will be calculated for each Group. The primary comparison will be Group R+AD vs. Group R and vs. Group AD | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Tom Smith, MD, Study Director — Teva Neuroscience, Inc.